CLINICAL TRIAL: NCT04888156
Title: Impact of Self-tonometry With iCare Home ® on Glaucoma Treatment Decision.
Brief Title: Impact of Self-tonometry on Glaucoma Treatment Decision.
Status: Completed | Type: Observational
Sponsor: St. Erik Eye Hospital (Other)
Responsible Party: Principal Investigator, Enping Chen, MD Ph D, St. Erik Eye Hospital
Other Study IDs: iCare Home
Record Dates: First submitted 2021-05-11; First posted 2021-05-17 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Glaucoma; Glaucoma, Open-Angle; OHT - Ocular Hypertension; Glaucoma Capsulare
Keywords: glaucoma; self-tonometry; treatment; IOP peaks
MeSH Terms: conditions — Glaucoma; Glaucoma, Open-Angle; Ocular Hypertension; Exfoliation Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GAT IOP below 15 mmHg: Glaucoma patients with an IOP measured with GAT below 15 mmHg prior performance of self-tonometry with iCare Home
  Interventions: Other: Unchanged treatment; Other: Changed treatment
- GAT IOP equal or above 15 mmHg: Glaucoma patients with an IOP measured with GAT equal or above 15 mmHg prior performance of self-tonometry with iCare Home
  Interventions: Other: Unchanged treatment; Other: Changed treatment

INTERVENTIONS:
Other: Unchanged treatment — Treatment is the same pre- and post self-tonometry
Other: Changed treatment — Treatment is changed post self-tonometry

SUMMARY:
Self-tonometry with iCare Home is performed by one hundred patients annually at Sankt Erik's Eye Hospital. The investigators want to evaluate the impact that self-tonometry results have on the clinician's choice of glaucoma treatment. The investigators also want to evaluate how often pressure peaks occur outside the clinic's opening hours.

DETAILED DESCRIPTION:
Since a few years back, self-tonometry has been available in glaucoma care. Self-tonometry allows patients to measure their eye pressure themselves using a portable tonometer. Sankt Erik's Eye Hospital was the first healthcare provider in Sweden to use this new technology. The investigators have previously conducted studies that have shown good agreement between the measurements made by patients and the gold standard method, e.g. Goldman applanation tonometry (GAT) (Chen, Querat et al. 2016, Querat and Chen 2017). About one hundred patients perform pressure curves with self-tonometry annually.

As the method is used regularly, the investigators want to evaluate the impact of self-tonometry results on the clinician's choice of glaucoma treatment. The investigators also want to evaluate how often pressure peaks occur outside the clinic's opening hours and how much they differ from GAT.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosed with POAG (primary open-angle glaucoma), PEX (pseudo-exfoliation glaucoma) or OHT (ocular hypertension)
* Difference between patients' and staff's iCare Home® measurements less than 5 mmHg at Baseline
* Difference between Goldman Applanation tonometry (GAT) and patient's highest iCare Home® measurements less than 7 mmHg at baseline
* Monitoring over at least two days

Exclusion Criteria:

* More than one measurement with iCare Home® tonometer below 5 mmHg
* Missing more than one daily measurement with iCare Home® tonometer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All glaucoma patients who obtained an IOP curve using an iCare Home® self-tonometer between January 2018 and December 2020 and who fulfill all the inclusion criteria and none of the exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Clinician's choice of glaucoma treatment | One month
  Type of treatment received by patient after performance of self-tonometry with iCare Home

SECONDARY OUTCOMES:
Occurence of IOP peaks | Three days of self-tonometry
  Occurence of IOP peaks measured by self-tonometry

CONTACTS AND LOCATIONS:
Overall Officials: Enping Chen, MD PhD, Principal Investigator — St. Erik Eye Hospital
Locations (1):
- St Erik Eye Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No